CLINICAL TRIAL: NCT03186677
Title: A Phase 1, Open-label, Multi-center, Dose-escalation Study to Investigate the Safety, Pharmacokinetics and Pharmacodynamics of ISU304 in Previously Treated Hemophilia B Patients
Brief Title: Dose-escalation Study to Investigate the Safety, PK, and PD of ISU304/CB2679d in Hemophilia B Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ISU Abxis Co., Ltd. (Industry)
Collaborators: Catalyst Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ISU304-001/CB2679d
Record Dates: First submitted 2017-05-30; First posted 2017-06-14 (Actual); Results first posted 2020-11-10 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-10

CONDITIONS: Hemophilia B
Keywords: ISU304; previously treated Hemophilia B patients; FIX; Factor IX; CB2679d; Dalcinonacog alfa
MeSH Terms: conditions — Hemophilia B | interventions — Factor IX

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Experimental): Single intravenous administration of BeneFIX (75 IU/kg) with 72 hours of observation, followed by single intravenous administration of ISU304/CB2679d/Dalcinonacog alfa (75 IU/kg) with 72 hours of observation
  Interventions: Biological: ISU304/CB2679d/Dalcinonacog alfa 75~150 IU/kg; Biological: BeneFIX
- Cohort 2 (Experimental): Single intravenous administration of ISU304/CB2679d/Dalcinonacog alfa (75 IU/kg) with 72 hours of observation, followed by single subcutaneous administration of ISU304/CB2679d/Dalcinonacog alfa (75 IU/kg) with 72 hours of observation
  Interventions: Biological: ISU304/CB2679d/Dalcinonacog alfa 75~150 IU/kg
- Cohort 3 (Experimental): Single intravenous administration of ISU304/CB2679d/Dalcinonacog alfa (75 IU/kg) with 72 hours of observation, followed by single subcutaneous administration of ISU304/CB2679d/Dalcinonacog alfa (150 IU/kg) with 120 hours of observation
  Interventions: Biological: ISU304/CB2679d/Dalcinonacog alfa 75~150 IU/kg
- Cohort 4 (Experimental): One subcutaneous administration of ISU304/CB2679d/Dalcinonacog alfa (150 IU/kg) per day for 6 days with 240 hours of observation
  Interventions: Biological: ISU304/CB2679d/Dalcinonacog alfa 75~150 IU/kg
- Cohort 5 (Experimental): One intravenous administration of ISU304/CB2679d/Dalcinonacog alfa (75 IU/kg) followed by subcutaneous administration of ISU304/CB2679d/Dalcinonacog alfa (150 IU/kg) once daily for 9 days with 312 hours of observation
  Interventions: Biological: ISU304/CB2679d/Dalcinonacog alfa 75~150 IU/kg

INTERVENTIONS:
Biological: ISU304/CB2679d/Dalcinonacog alfa 75~150 IU/kg — ISU304/CB2679d/Dalcinonacog alfa 75~150 IU/kg by intravenous or subcutaneous
  Other Names: Dalcinonacog alfa
Biological: BeneFIX — BeneFIX 75 IU/kg, intravenous administration
  Arms: Cohort 1

SUMMARY:
This study is a phase 1, open-label, multi-center, dose-escalation study to investigate the safety, pharmacokinetics and pharmacodynamics of ISU304/CB2679d in previously treated hemophilia B patients.

DETAILED DESCRIPTION:
This study is a phase 1, open-label, multi-center, dose-escalation study to investigate the safety, pharmacokinetics, and pharmacodynamics of ISU304/CB2679d/Dalcinonacog alfa in previously treated Hemophilia B patients.

This study is comprised of 5 cohorts. Each cohort may receive an intravenous administration of 75 IU/kg, with subcutaneous administrations from 75 IU/kg to 150 IU/kg.

During the study period, a subject may be hospitalized to facilitate the collection of blood samples for pharmacokinetic (PK)/pharmacodynamic (PD) analysis. The Data Safety Monitoring Board (DSMB) and Data Monitoring Committee (DMC) will be operated after the end of Cohorts 1 to 4. These committees will monitor the PK/PD and safety data from each cohort to determine the continuation of next cohort (Cohorts 2 to 5), target dose, and blood sampling period for PK/PD (including timing of collection). Additional subjects may be enrolled in all cohorts or cohorts may be canceled depending on the results of PK/PD analysis. A cohort of subcutaneous dosing at 300 IU/kg was cancelled as single-dose PK is uninformative.

ELIGIBILITY:
Inclusion Criteria:

1. Previously treated male patients with moderate or severe hemophilia B (documented FIX activity ≤ 2% and exposed to any FIX product for ≥ 150 exposure days (estimated) at the time of screening)
2. Patients must be 12 to 65 years old at the time of screening
3. Patients who have discontinued a previously treated FIX product at least 4 days prior to the administration of investigational product
4. HIV negative, or if HIV positive with a CD4 count > 200/μL (documented < 200 particles/μL or ≤ 400,000 copies/mL) at the time of screening
5. Voluntary consent to participate in the study

Exclusion Criteria:

1. Patients with a history or a family history of FIX inhibitors
2. Patients with FIX inhibitors (positive result for BeneFIX or ISU304 from inhibitor tests) at the time of screening
3. Patients who have a history of thromboembolic events (myocardial infarction, cerebrovascular disease, venous thrombosis, etc.)
4. Patients with known hypersensitivity, allergy, or anaphylaxis to any FIX product or hamster protein
5. Patients receiving treatment with a FIX product or a bypass agent within 4 half-lives for the agent used (at least 96 hours) prior to the administration of the investigational product
6. Patients who have been exposed to long-term administration of immunomodulating agents or immunosuppressants such as α-INF or adrenocortical hormones over the past 3 months or who are currently receiving or planning to receive such treatment during the study period
7. Patients who have been administered vaccines during the period of 6 months prior to the administration of the investigational product or plan to receive vaccines during the study period
8. Patients with any other co-existing bleeding disorder (Von Willebrand disease, etc.)
9. Patients with positive D-dimer results (≥ 0.5 μg/mL) at the time of screening
10. Patients with platelet counts less than 100,000/μL at the time of screening
11. Patients with ALT, AST levels 5 times greater than upper normal limit or total bilirubin, serum creatinine levels 2 times greater than upper normal limit at the time of screening
12. Active hepatitis patients who are HBs Ag positive or anti-HCV Ab positive at the time of screening
13. Patients scheduled for surgery during the study period
14. Patients participated in another study within 30 days before screening or scheduled to participate in any other study during the study period

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-06-03 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2019-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ChurWoo You, PhD, Principal Investigator — Eulji University Hospital Seo-gu
Locations (3):
- South Korea (3):
  - Eulji University Hospital, Daejeon
  - Pusan National Univesity Hospital, Pusan
  - Yonsei University Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Faraj A, Le Moan N, Gorina E, Blouse GE, Knudsen T, Simonsson USH. Model-Informed Support of Dose Selection for Prophylactic Treatment with Dalcinonacog Alfa in Adult and Paediatric Hemophilia B Patients. Adv Ther. 2023 Sep;40(9):3739-3750. doi: 10.1007/s12325-023-02570-6. Epub 2023 Jun 21. PMID 37341915

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 11 unique subjects who completed the study; 2 failed screening. Of the 5 subjects in Cohort 4, 1 subject previously participated in Cohort 1 and 2 subjects in Cohort 2. Of the 2 subjects in Cohort 5, 2 subjects previously participated in Cohort 4. As a result, the Safety Analysis Set included 16 subjects. Cohorts were conducted in numerical order.
Groups:
- Period 1, Cohort 1: Single intravenous administration of BeneFIX (75 IU/kg) with 72 hours of observation, followed by single intravenous administration of ISU304/CB2679d/Dalcinonacog alfa (75 IU/kg) with 72 hours of observation
- Period 1, Cohort 2: Single intravenous administration of ISU304/CB2679d/Dalcinonacog alfa (75 IU/kg) with 72 hours of observation, followed by single subcutaneous administration of ISU304/CB2679d/Dalcinonacog alfa (75 IU/kg) with 72 hours of observation
- Period 1, Cohort 3: Single intravenous administration of ISU304/CB2679d/Dalcinonacog alfa (75 IU/kg) with 72 hours of observation, followed by single subcutaneous administration of ISU304/CB2679d/Dalcinonacog alfa (150 IU/kg) with 120 hours of observation
- Period 2, Cohort 4: One subcutaneous administration of ISU304/CB2679d/Dalcinonacog alfa (150 IU/kg) per day for 6 days with 240 hours of observation
- Period 2, Cohort 5: One intravenous administration of ISU304/CB2679d/Dalcinonacog alfa (75 IU/kg) followed by subcutaneous administration of ISU304/CB2679d/Dalcinonacog alfa (150 IU/kg) once daily for 9 days with 312 hours of observation
Period: Period 1
Arm/Group | Period 1, Cohort 1 | Period 1, Cohort 2 | Period 1, Cohort 3 | Period 2, Cohort 4 | Period 2, Cohort 5
Started | 3 | 3 | 3 | 0 | 0
Completed | 3 | 3 | 3 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Period 1, Cohort 1 | Period 1, Cohort 2 | Period 1, Cohort 3 | Period 2, Cohort 4 | Period 2, Cohort 5
Started | 0 | 0 | 0 | 5 | 2
Completed | 0 | 0 | 0 | 5 | 2
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: There were 13 unique subjects in the study: 11 completed study and 2 failed screening. Of the 11 individuals who completed the study, 5 were in multiple cohorts. Baseline characteristics are reported according to the initial cohort to which subjects were assigned. The 2 subjects who participated in Cohort 5 were previously in Cohort 4.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Total
Number analyzed (Participants) | 3 | 3 | 3 | 2 | 0 | 11
Age, Categorical [Count of Participants; unit: Participants] — Population: There were 13 unique subjects in the study; 11 completed study and 2 failed screening. Of the 11 individuals who completed the study, 5 were in multiple cohorts. 16 subjects were included in the Safety Analysis Set across 5 cohorts.
  Participants
    <=18 years | 1 | 0 | 0 | 0 | 0 | 1
    Between 18 and 65 years | 2 | 3 | 3 | 2 | 0 | 10
    >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.00 (16.70) | 46.33 (5.69) | 43.33 (14.57) | 50.50 (3.87) |  | 41.55 (13.68)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: There were 13 unique subjects in the study; 11 completed study and 2 failed screening. Of the 11 individuals who completed the study, 5 were in multiple cohorts. 16 subjects were included in the Safety Analysis Set across 5 cohorts.
  Participants
    Female | 0 | 0 | 0 | 0 | 0 | 0
    Male | 3 | 3 | 3 | 2 | 0 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 3 | 3 | 2 | 0 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 3 | 3 | 3 | 2 | 0 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events (AEs) After the Administration of Investigational Products (IP)
Description: The number of reported AEs (local/systemic/other) after IP administration was calculated by cohort.
Time Frame: Through study completion, an average of 8 days
Population: There were 13 unique subjects in the study: 11 completed study and 2 failed screening. Of the 11 individuals who completed the study, 5 were in multiple cohorts. 16 subjects were included in the Safety Analysis Set across 5 cohorts.
Measure: Number; unit: adverse events
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 3 | 3 | 3 | 5 | 2
adverse events | 0 | 10 | 10 | 69 | 47

2. Secondary Outcome: Maximum Plasma Concentration (Cmax)
Description: Cmax analysis was conducted by cohort as a Factor IX (FIX) potency percent
Time Frame: 0 to 72 hours for Cohorts 1 to 3, 0 to 120 hours for Cohorts 4 and 5
Measure: Mean (Standard Deviation); unit: FIX potency percent
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 3 | 3 | 3 | 5 | 2
FIX potency percent
  Cmax of ISU304/CB2679d/Dalcinonacog alfa IV | 71.10 (15.87) | 100.80 (78.00) | 41.70 (7.47) | 15.34 (2.44) | 23.80 (10.04)
  Cmax of ISU304/CB2679d/Dalcinonacog alfa SC | 70.47 (16.92) | 5.30 (3.69) | 5.27 (1.16) | NA (NA) — Cmax calculated for only one treatment and route of administration (subcutaneous) in this cohort. | NA (NA) — Cmax calculated for only one treatment and route of administration (subcutaneous) in this cohort.

3. Secondary Outcome: Factor IX Inhibitor
Description: The presence/absence of Factor IX (FIX) neutralizing antibodies was assessed by ELISA anti-drug assay [Dalcinonacog alfa and BeneFIX) and if positive, a modified Nijmegen assay for each subject by cohort at end of study visit.
  Measure description: count of participants with neutralizing antibodies. Bethesda Units >0.6 indicates presence of neutralizing antibodies. 1 BU is defined as a 50% reduction in FIX activity when adding participant plasma to a standard with known FIX activity.
Time Frame: At end of study visit (an average of 8 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 3 | 3 | 3 | 5 | 2
Participants | 0 | 0 | 0 | 0 | 2

ADVERSE EVENTS:
Time Frame: For 7 to 15 days depending on the cohort: Cohort 1 (7 days), Cohort 2 (7 days), Cohort 3 (9 days), Cohort 4 (10 days), Cohort 5 (15 days)
Groups:
- Cohort 5: One intravenous administration of ISU304/CB2679d/Dalcinonacog alfa (75 IU/kg) followed subcutaneous administration of ISU304/CB2679d/Dalcinonacog alfa (150 IU/kg) once daily for 9 days with 312 hours of observation
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/5 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/5 | 0/2
Other Adverse Events (participants affected / at risk) | 0/3 | 3/3 | 3/3 | 5/5 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=3) | Cohort 3 (N=3) | Cohort 4 (N=5) | Cohort 5 (N=2)
Injection site pain (General disorders) | 0 (0) | 2 (2) | 3 (3) | 5 (34) | 2 (11)
Injection site erythema (General disorders) | 0 (0) | 1 (2) | 3 (3) | 2 (32) | 2 (15)
Injection site papule (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (9)
Injection site pruritus (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Injection site discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anti ISU304 antibody positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)

LIMITATIONS AND CAVEATS:
Two subjects who were cousins developed neutralizing antibodies to dalcinonacog alfa in Cohort 5 that did not cross react with wild-type FIX. Both resumed their prior FIX therapy. Five subjects participated in 2 cohorts each.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-11): https://cdn.clinicaltrials.gov/large-docs/77/NCT03186677/Prot_SAP_000.pdf